Statistical analysis plan.

Study name: The use of Focused Lung Ultrasound in Patients Suspected of COVID-19.

## 8.April 2020

| Descriptive data: | | |
|-------------------|------------------|-----------|
| Demographic | Age | Mean, sd |
| | Sex | % kvinder |
| | Weight | Mean, sd. |
| | Height | Mean, sd. |
| | Site | groupe |
| Baseline data | BT sys | Mean, sd. |
| | BT dia | Mean, sd. |
| | SAT | Mean, sd. |
| | Puls | Mean, sd. |
| | Respiratory Rate | Mean, sd. |
| | Oxygen, I/min | Mean, sd. |
| | ferritin | Mean, sd. |
| | Hbg | Mean, sd. |
| | Leukocytter | Mean, sd. |
| | Lymfocytter | Mean, sd. |
| | Mono | Mean, sd. |
| | Neutrofile | Mean, sd. |
| | Egfr | Mean, sd. |
| | Karbamid | Mean, sd. |
| | Kreatinin | Mean, sd. |
| | Natrum | Mean, sd. |
| | Kalium | Mean, sd. |
| | Ddimer | Mean, sd. |
| | Probnp | Mean, sd. |
| | Tnt | Mean, sd. |
| | Tni | Mean, sd. |
| | glucose hba1c | Mean, sd. |
| | ph | Mean, sd. |
| | pco2 | Mean, sd. |
| | po2 | Mean, sd. |
| | be | Mean, sd. |
| | bicarbonat | Mean, sd. |
| | lactat | Mean, sd. |
| | Rtg af thorax | Grupper |
| | CT thorax | Grupper |
| | Covid-19 pcr | Yes/No |
| Treatment data | Antibiotica | Yes/No |
| | Antiviral | Yes/No |

| | | Biological | Yes/No | |
|---|---|---|---|---|
| | | Anti thormbotic | Yes/No | |
| | | | Yes/No | |
| | | Death during admission | 163/110 | |
| | | Length of | kontinuert | |
| | | admission | Kontinuert | |
| | | | Voc/No | |
| | | Death at 30 days Cause of death | Yes/No | |
| | | | Covid/ikke-covid | |
| | | Treatment | Yes/No | |
| | | restrictions, ITA | /NI - | |
| | | Treatment | Yes/No | |
| | | restrictions, | | |
| = | | ventilator | | |
| FLUS data. | | L1 | 0-3 | |
| | | L2 | 0-3 | |
| | | L3 | 0-3 | |
| | | L4 | 0-3 | |
| | | L5 | 0-3 | |
| | | L6 | 0-3 | |
| | | L7 | 0-3 | |
| | | R1 | 0-3 | |
| | | R2 | 0-3 | |
| | | R3 | 0-3 | |
| | | R4 | 0-3 | |
| | | | 0-3 | |
| | | R6 | 0-3 | |
| | | | 0-3 | |
| | | Flus mean | 0-3, sd | |
| Inter- intraobser | vatør agreement | | | |
| Limits of agreemen | | 20% Flus film re- | Weigthed kappa | kap s1 s2, tab |
| Bland altmann. | | scored by | | wgt(w) |
| Diana aidinanii. | | 1.observatør | | **BC(**) |
| | | 20% Flus film | Weigthed kappa | kap o1 o2, tab |
| | | scored by | **Ciguica kappa | wgt(w) |
| | | 2.observatør | | **S(\**) |
| Moan Flue sooms | rolatored tal aver | - L | | |
| | relatered tol ever | | | |
| Covid death | Parametric destribution qq plot and histogram | | | |
| | Norm + | t-test. | ttest flusmed, by(cov | |
| | Nomr - | Wilcoxon | ranksum flusmed, by | (covdod) |
| | | | by covdod, sort : summarize flusmed, d | |
| ITA l | graph bar (Mean) flusmed, over(covdod) | | | |
| ITA admission | Parametric destribution qq plot and histogram | | | |
| | Norm + | t-test. | ttest flusmed, by(ita_in) | |
| | Nomr - | Wilcoxon | by ita_in, sort : summarize flusmed, d | |
| | | | | /·· · · · |
| | | | ranksum flusmed, by | (ıta_in) |

| | | | graph bar (Mean) flusmed, over(ita_in) |
|---|---|---|---|
| Ventilator<br>treatment | Parametric destribution qq plot and histogram | | |
| | Norm + | t-test. | ttest flusmed, by(respirator_beh) |
| | Nomr - | Wilcoxon | by respirator_beh, sort : summarize flusmed, d ranksum flusmed, by(respirator_beh) graph bar (Mean) flusmed, over(respirator_beh) |
| Prædiction of e | event | | |
| Covid death | Univariat logistical regression | Variable: covdod flusmed | |
| | Multivariate<br>logistical<br>regression | Variable: covdod,<br>Flusmed, alder,<br>køn, sat, ilt<br>(kategori?) | |
| ITA admission | Univariat<br>logistiscal<br>regression | Variable: ita_in<br>flusmed | |
| | Multivariate logistical regression | Variable: ita_in,<br>Flusmed, alder,<br>køn, sat | , if behandlingsloft_ita ==0 |
| Ventilator<br>treatment | Univariat logistical regression | Variable:<br>respirator_beh<br>flusmed | |
| | Multivariate<br>logistical<br>regression | Variable:<br>respirator_beh<br>Flusmed, alder,<br>køn, sat | , if behandlingsloft_resp ==0 |

Continuous variables are assessed for parametric distribution with quartile-quartile plots. Medians, interquartile ranges or means and standard deviations and ranges are reported according to parametric distribution. Students' t-test or Mann-Whitney U test is used as it was considered appropriate to evaluate differences between groups. The statistical significance is set to 5%. All data are handled in Excel (Microsoft) and REDCap (hosted at Aarhus University). All analyses are performed using Stata 14.2 (StataCorp, USA).

## **Building Prediction Models**

Prediction models are based on multivariable logistic regression and preselected variables. The variables are sex, age, relevant comorbidity, oxygen administration and the mean-FLUS score. The selection of these variables is based on published data and clinical experience available to the study group during the study design stage. Explanatory variables are examined to decide cut-points, scales or the need for transformation. Variables are limited and prioritized to avoid overfitting or underfitting, respecting the study population size. Every included variable require at least 15 events.

The dependent variable is the primary outcome of interest: the COVID-19-related need for mechanical ventilation in the main analysis. Secondary outcomes are analyzed using the same logistic regression model, except for the outcome on high-flow oxygen treatment. The explanatory variable on oxygen administration is considered closely related to the outcome and is thus excluded from this analysis.